CLINICAL TRIAL: NCT01623518
Title: A Phase I Study to Determine the Safety and Immunogenicity of the Candidate Influenza Vaccine ChAdOx1-NP+M1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FLU004; 2012-000641-12 (EudraCT Number)
Record Dates: First submitted 2012-06-13; First posted 2012-06-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ChAdOx1-NP+M1 (Experimental)
  Interventions: Biological: ChAdOx1-NP+M1

INTERVENTIONS:
Biological: ChAdOx1-NP+M1 — Dose escalation in a 3+3 study plan;
  5 x10^8 vp, 5 x10^9 vp, 2.5 x10^10 vp, 5 x10^10 vp

SUMMARY:
This is a first in man dose escalation study, to assess the safety and immunogenicity of the candidate influenza vaccine ChAdOx1-NP+M1. All volunteers recruited will be healthy adults aged 18-50. Volunteers will be enrolled and doses will be escalated according to a "3+3" study plan. Up to 24 volunteers will be vaccinated. Following one dose of the vaccine, volunteers will be followed up to assess the side effect profile of the vaccine and to take blood tests. A series of immunology assays will be performed to determine how potent the vaccine is at inducing an immune response.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Men and women aged 18-50
* Resident in or near Oxford for the duration of the vaccination study
* Able and willing (in the Investigators' opinions) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* Willingness to use effective contraception for 4 weeks from the date of vaccination
* Agreement to refrain from blood donation for 4 weeks from the date of vaccination
* Written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Previous receipt of any recombinant adenoviral vectored vaccine
* Previous receipt of MVA-NP+M1
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled/topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis in reaction to vaccination
* History of cancer (except basal cell carcinoma and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any chronic illness requiring ongoing or awaiting hospital specialist supervision, other than minor surgical procedures and follow up of surgery over 6 months prior to screening.
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface (HBsAg) or hepatitis C virus (antibodies to HCV)
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigators, would either put the volunteer at risk because of participation in the study, or may influence the result of the study.
* No response / confirmation from GP regarding previous medical history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety | 3 weeks
  Analysis of data on adverse events.

SECONDARY OUTCOMES:
Reactogenicity | 3 weeks
  Immunogenicity endpoints will include interferon-gamma ELISpot as a marker of cell-mediated immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hill, MD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom